## **ANNEX: INFORMED CONSENT (TRANSLATION TO ENGLISH)**



Date:

| PATIENT CONSENT |
|---|
| (Biomedical Investigation Law 14/2007) |
| (Data protection Law 3/2018) |
| (Data protection general ruling 2016/679) |
| (Patient autonomy law 41/2002) |
| STUDY TITLE: "VIDEO DISCHARGE INSTRUCTIONS FOR PEDIATRIC GASTROENTERITIS IN AN EMERGENCY DEPARTMENT: A RANDOMIZED, CONTROLLED TRIAL" |
| Código: GEA01<br>Versión: 1.2 (English versión) |
| Rafael Marañón Pardillo. Pediatric Emergency Department. 91 529 01 72 |
| Ana Jové Blanco. Pediatric Emergency Department. 91 529 01 72 |
| Gonzalo Solís García. Pediatric Emergency Department. 91 529 01 72 |
| CENTER: Hospital General Universitario Gregorio Marañón. |
| I,, declare under my own responsibility that I have read the Information Sheet about the study and voluntarily accept participating. |
| 2. I have been given a copy of the Information Sheet and a copy of Informed Consent, dated and signed. I have been information about characteristics and aim of the study, and about the possible benefits and risks associated to it. I have been given time and opportunity to pose questions. All asked questions |
| were properly answered. 3. I know that identities of subjects participating will be kept in secret and will be identified with a purposited gode. |
| <ul><li>identified with a numerical code.</li><li>4. I am free to retire from the study at any time and for any reason, without giving any explanation and without repercussions in my future medical treatment</li></ul> |
| 5. I understand that the aim of the study Is to evaluate the population included and<br>that the results will not be communicated to me nor my doctor, unless the<br>results have a significant importance in the patients' health and there is a real<br>possibility to improve your health. |
| Point 1 I VOLUNTARILY GIVE my consent for this study. |
| Point 2 I VOLUNTARILY GIVE my consent for my data to be kept anonymously. |

Parent or tutor sign:

| I declare | e that I have | explained th | e characteri | ristics and a | im of the | study, 1 | the dif | ferent |
|---|---|---|---|---|---|---|---|---|
| parts and the p | otential bene | fits and risks | s, to the su | bject which | signs this | form. | The p | atient |
| consents participating in this study by signing and dating this document. | | | | | | | | |

Signo of the Investigator

| CANCELLING OF INFORMED CONS | SENT |
|---|---|
| I, with date | _, cancel the informed consent for participating in this study. |
| Caregiver or tutor Sign | Sign of the investigator |